CLINICAL TRIAL: NCT00850954
Title: Project CASA: Promoting Smoke-Free Indoor Air Policy in Mexican American Households
Brief Title: Project CASA in Promoting Smoke-Free Indoor Air Policy in Mexican American Households
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2006-0440; NCI-2019-02502 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006-0440 (Other: M D Anderson Cancer Center); P30CA016672 (NIH)
Record Dates: First submitted 2009-02-24; First posted 2009-02-25 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2022-06

CONDITIONS: Cigarette Smoker; Current Smoker; Currently Living With Smoker
MeSH Terms: interventions — Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (smoking cessation) (Experimental): Participants receive smoking cessation intervention materials based on TTM.
  Interventions: Behavioral: Smoking Cessation Intervention; Other: Survey Administration
- Group II (informational) (Experimental): Participants receive fotonovelas and other materials on secondhand smoking and how to assist the smoker in quitting.
  Interventions: Other: Informational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Informational Intervention — Receive information on secondhand smoke and supporting smoker in quitting
  Arms: Group II (informational)
Behavioral: Smoking Cessation Intervention — Receive smoking cessation materials based on TTM
  Other Names: Smoking and Tobacco Use Cessation Interventions
  Arms: Group I (smoking cessation)
Other: Survey Administration — Ancillary studies

SUMMARY:
This trial studies the effect of an intervention program, Project CASA, on smoking cessation and reducing secondhand smoke exposure in Mexican American households. Project CASA, comprising pamphlets and fotonovelas (illustrated storybooks), may provide valuable information to participants on how to improve the air quality in their homes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Reduction in secondhand smoke exposure: The study will distinguish if a tailored intervention designed to address the needs of the target group will reduce objectively and subjectively measured secondhand smoke exposure of nonsmokers in Mexican American (MA) households.

Ia. Develop tailored fotonovelas for intervention implementation. II. Smoking cessation: The study will identify if a tailored intervention designed to address the needs of the target group will help the primary smokers in the household quit smoking.

III. Stages of change: The study will identify if the proposed intervention will have a significant impact on the primary smoker(s) progression through the stages of smoking cessation.

IV. Knowledge and attitudes: The study will identify if the proposed intervention will result in better knowledge and changed attitudes towards secondhand smoke exposure among members of MA households (smokers and nonsmokers) compared to standard care.

V. Perceived health: The study will distinguish whether reduced exposure to secondhand smoke would improve perceived health.

OUTLINE: Participants are assigned to 1 of 2 groups based on smoking status.

GROUP I (SMOKERS): Participants receive smoking cessation intervention materials based on transtheoretical model of change (TTM).

GROUP II (NON-SMOKERS): Participants receive fotonovelas and other materials on secondhand smoking and how to assist the smoker in quitting.

Participants are followed up at 6 and 12 months to assess for home air quality.

ELIGIBILITY:
Inclusion Criteria:

* Live in the targeted Mexican American neighborhoods.
* Can read Fotonovelas in English and Spanish.
* Access to telephone.
* Smoker in household (adult [18+] person living in the household who smokes INSIDE at least one cigarette a week).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2006-08-08 (Actual); Primary Completion 2018-08-07 (Actual); Study Completion 2018-08-07 (Actual)

PRIMARY OUTCOMES:
Level of nicotine measured at 6 month post intervention | 6 months after treatment
  Method of analysis is a pre-post test analysis of covariance, ANCOVA, using a linear regression model (PROC REG in SAS). In this analysis, the prevalence of nicotine levels at the 6-month follow-up compared between conditions while controlling for baseline nicotine levels. Second hand smoke (SHS) exposure based on objective monitoring of SHS in each household (in the kitchen and TV room) over a 7-day period. A small, lightweight (16 gram) passive nicotine monitor used to measure exposure to nicotine.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Prokhorov, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org